CLINICAL TRIAL: NCT00265343
Title: A Multicenter, Double-Blind, Flexible-Dose, 6-Month Extension Trial Comparing the Safety and Efficacy of Asenapine With Olanzapine in Subjects Who Completed the Protocol 25543 (NCT 00212836; P05817)
Brief Title: 6-Month Extension Trial of Asenapine With Olanzapine in Negative Symptom Patients Who Completed the Protocol 25543 (25544)(P05777)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05777; 25544; Aphrodite
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): asenapine
  Interventions: Drug: asenapine
- 2 (Active Comparator): olanzapine
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — 5-10 mg sublingually twice daily for 26 weeks
  Arms: 1
Drug: olanzapine — 5-20 mg by mouth once daily for 26 weeks
  Arms: 2

SUMMARY:
This is an extension study to further test

the efficacy and safety of asenapine compared with a

marketed agent (olanzapine) in the treatment of patients with

persistent negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Continue to meet all demographic and procedural

inclusion criteria of the 25543 trial (NCT 00212836; P05817) to enter into

this extension trial.

* Have demonstrated an acceptable

degree of compliance and completed the 25543

trial, and would benefit from continued treatment

according to the investigator.

Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant

medical condition.

* Have been judged to be medically

noncompliant in the management of their disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Result] Buchanan RW, Panagides J, Zhao J, Phiri P, den Hollander W, Ha X, Kouassi A, Alphs L, Schooler N, Szegedi A, Cazorla P. Asenapine versus olanzapine in people with persistent negative symptoms of schizophrenia. J Clin Psychopharmacol. 2012 Feb;32(1):36-45. doi: 10.1097/JCP.0b013e31823f880a. PMID 22198451

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine: 5-10 mg twice daily (bid) sublingual (SL)
- Olanzapine: 5-20 mg daily (QD) orally (PO)
Period: Overall Study
Arm/Group | Asenapine | Olanzapine
Started | 134 | 172
Completed | 113 | 153
Not Completed | 21 | 19
Not completed — Adverse Event | 10 | 7
Not completed — Withdrawal by Subject | 3 | 9
Not completed — Other | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine | Olanzapine | Total
Number analyzed (Participants) | 134 | 172 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.2) | 40.7 (11.7) | 40.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 53 | 96
  Male | 91 | 119 | 210

OUTCOME MEASURES:

1. Primary Outcome: Long-term Change in Negative Symptoms of Schizophrenia Measured by the Negative Symptom Assessment (NSA) Scale
Description: Decrease from baseline in the NSA scores indicates improvement of efficacy. Range NSA total score is 16 [best]-96 [worst].
Time Frame: Baseline of Protocol 25543 (NCT 00212836) to 365 days (total time for both protocols 25543 & 25544)
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 122 | 157
Units on a Scale | -16.9 (0.98) | -15.4 (0.85)

2. Secondary Outcome: Change in Quality of Life Measured by Quality of Life Scale (QLS)
Description: Increase from baseline in the QLS scores indicates improvement of efficacy. Range QLS total score is 0 [worst]-126 [best].
Time Frame: Baseline of Protocol 25543 (NCT 00212836) to 365 days (total time for both protocols 25543 & 25544)
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 122 | 157
Units on a Scale | 18.7 (1.64) | 16.4 (1.4)

ADVERSE EVENTS:
Arm/Group | Asenapine | Olanzapine
Serious Adverse Events (participants affected / at risk) | 9/134 | 6/172
Other Adverse Events (participants affected / at risk) | 19/134 | 21/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=134) | Olanzapine (N=172)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (3) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 4 (4) | 3 (3)
Stress (Psychiatric disorders) | 1 (3) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=134) | Olanzapine (N=172)
Influenza (Infections and infestations) | 7 (7) | 3 (3)
Weight increased (Investigations) | 0 (0) | 11 (11)
Headache (Nervous system disorders) | 7 (8) | 7 (8)
Schizophrenia (Psychiatric disorders) | 7 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication/presentation of data may not be made without prior review and comment by the Sponsor; all reasonable comments of Sponsor will be incorporated as far as the scientific data content is not impaired. A complete copy shall be provided to the Sponsor at least 60 days prior to date of submission. Participation in the Study involves a commitment to publish data from the study in a cooperative publication prior to publication/presentation or on an individual basis.